CLINICAL TRIAL: NCT06890806
Title: Comparison of the Effects of Foot Core Stabilization Exercises Versus Extracorporeal Shock Wave Therapy (ESWT) on Pain, Muscle Strength and Functionality in Individuals with Plantar Fasciitis
Brief Title: Foot Core Stabilization Exercises Vs. Shockwave Therapy for Pain, Strength, and Function in Plantar Fasciitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gulay karacaoglu, asisstant prof., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-7450
Record Dates: First submitted 2025-03-11; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Plantar Fasciitis of Both Feet
Keywords: Extracorporeal Shock Wave Therapy; Pain; Foot stabilization exercises
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The participants will be divided into two groups for treatment. One group will receive extracorporeal shock wave therapy (ESWT), while the other group will undergo stabilization exercises.
Who Masked: Participant
Masking Description: The participants were unaware of which group they would be assigned to. Based on the order of their arrival at the hospital, those who came in first, third, fifth, etc., were assigned to the Extracorporeal Shock Wave Therapy (ESWT) group, while those who came in second, fourth, sixth, etc., were assigned to the Stabilization Exercises group. This allocation method ensured that participants remained blinded to their group assignment, minimizing potential bias in their responses or expectations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foot Core Stabilization Exercise Group (FCSEG) (Experimental): Foot Core Stabilization Exercise Group (FCSEG)
  Interventions: Other: Foot Core Stabilization Exercise Group (FCSEG)
- Extracorporeal Shock Wave Therapy Group (ESWTG) (Experimental): Extracorporeal Shock Wave Therapy Group (ESWTG)
  Interventions: Other: Extracorporeal Shock Wave Therapy Group (ESWTG)

INTERVENTIONS:
Other: Foot Core Stabilization Exercise Group (FCSEG) — Exercise Group (Foot Core Stabilization Exercises)
  Exercise Group will perform foot core stabilization exercises under the supervision of a physiotherapist, three times a week for five weeks. The exercises will include:
  Short foot exercise Towel curl exercise Big toe press exercise Toe splay exercise Calf raise to big toe press exercise Leg swings Backward tandem walking Each exercise will be performed in three sets of 15 repetitions.
  Arms: Foot Core Stabilization Exercise Group (FCSEG)
Other: Extracorporeal Shock Wave Therapy Group (ESWTG) — Extracorporeal Shock Wave Therapy Group (ESWTG) One group will receive Extracorporeal Shock Wave Therapy (ESWT) once a week for five weeks. The ESWT sessions will be performed using the Gymna Shockmaster 500 device at a frequency of 15 Hz and a pressure of 3 bar, delivering a total of 1800 pulses per session.
  Arms: Extracorporeal Shock Wave Therapy Group (ESWTG)

SUMMARY:
This study aims to evaluate the effectiveness and feasibility of two distinct approache extracorporeal shock wave therapy and foot core stabilization exercises in the treatment of plantar faciitis (PF) by comparing their impacts on pain, muscle strength, and functionality. The study seeks to better understand the role of innovative exercise protocols in addressing biomechanical imbalances and the contribution of ESWT to biological healing mechanisms. The anticipated results are expected to provide evidence-based treatment approaches that can enhance the quality of life in individuals with PF, guide clinical applications in physical medicine and rehabilitation, and strengthen the position of these treatment methods within the broader healthcare system. Moreover, the findings may benefit a larger patient population by improving the management of PF.

DETAILED DESCRIPTION:
Participants aged 25-60 years who applied to the Physical Medicine and Rehabilitation Department of Bursa VM Medical Park Hospital and were diagnosed with plantar fasciitis (PF) by a physical medicine and rehabilitation physician or orthopedist will be included in the study. A total of 40 participants will be randomized, with 20 individuals in each group. Randomization will be based on the order of participant enrollment. The groups will be named the Foot Core Stabilization Exercise Group (ACSEG) and the Extracorporeal Shock Wave Therapy Group (ESWTG).

Informed consent forms will be obtained from individuals who meet the inclusion criteria. After collecting sociodemographic information, the following assessment methods will be applied, and the results will be recorded in the pre- and post-treatment evaluation form.

Evaluation:

After collecting sociodemographic information, participants' pain will be assessed using the Visual Analog Scale (VAS), medial longitudinal arch (MLA) height will be evaluated using the Navicular Drop Test, muscle strength will be measured using the Kinvent K-Force device, the relationship between foot structure and lower extremity biomechanics will be assessed using the Quadriceps (Q) Angle measured with a goniometer, foot posture will be evaluated using the Foot Posture Index (FPI), and foot function will be assessed using the Foot Function Index (FFI). All evaluations will be conducted under the supervision of an expert physiotherapist.

Sociodemographic Information:

The names, ages, heights, weights, body mass indices (BMI), and occupations of the participants with PF will be recorded.

Visual Analog Scale (VAS):

The VAS will be used to assess heel pain in individuals with PF. Participants will mark their pain on a 10 cm scale, where 0 represents no pain and 10 represents severe pain.

Navicular Drop Test:

The Navicular Drop Test will be used to evaluate MLA height. The navicular tubercle will be marked with a pen while the participant stands barefoot. The distance between the navicular tubercle and the ground will be measured in millimeters (mm) while the participant is seated without bearing weight on the foot. The participant will then stand and bear full weight on the foot, and the distance will be measured again. The difference between the two measurements will be recorded. Results will be classified as increased supination (<5 mm), neutral foot (5-9 mm), or increased pronation (>9 mm).

Muscle Strength Measurement:

Muscle strength will be measured using the Kinvent K-Force device. Participants will lie supine, and the dynamometer will be placed on the upper metatarsal region for dorsiflexor strength and the plantar metatarsal region for plantar flexor strength. Participants will push against the dynamometer with maximum force, and the results will be recorded.

Quadriceps (Q) Angle Measurement:

The Q angle will be measured using a plastic goniometer. Participants will lie supine with their knees extended. The goniometer's pivot point will be placed at the midpoint of the patella, with the movable arm pointing to the anterior superior iliac spine and the fixed arm aligned with the tibial tuberosity. The angle between the two arms will be recorded as the Q angle.

Foot Posture Index (FPI):

Foot posture will be assessed using the Foot Posture Index. Participants will stand in a relaxed position, looking forward, with arms at their sides and maintaining proper body alignment. Six clinical criteria will be evaluated:

Palpation of the talar head. Curves above and below the lateral malleolus. Inversion/eversion of the calcaneus. Bulging in the talonavicular joint region. Structure of the MLA. Forefoot abduction/adduction relative to the hindfoot. Each criterion will be scored from -2 to +2, with the total score recorded. A score of 0 indicates a neutral foot, positive values indicate pronation, and negative values indicate supination.

Foot Function Index (FFI):

The FFI evaluates foot pain, disability, and activity limitations through 23 items divided into three subscales. The pain subscale measures the level of foot pain in various situations, the disability subscale assesses the difficulty of performing functional activities due to foot problems, and the activity limitation subscale evaluates restrictions caused by foot problems. Participants will score each item based on their foot condition over the past week using the VAS.

Treatment:

The Foot Core Stabilization Exercise Group (ACSEG) will receive foot core stabilization exercises, while the Extracorporeal Shock Wave Therapy Group (ESWTG) will undergo shock wave therapy.

Extracorporeal Shock Wave Therapy Group (ESWTG):

ESWT will be administered using the Gymna Shockmaster 500 device by an expert physiotherapist. The therapy will be applied in continuous mode at 15 Hz frequency, with a pressure of 3 bars, delivering 1800 pulses per session. Treatment will be administered once a week for five weeks. After identifying the painful area on the heel, 200 pulses will be applied to each of the nine points, totaling 1800 pulses.

Foot Core Stabilization Exercise Group (ACSEG):

Participants will perform foot core stabilization exercises under the supervision of an expert physiotherapist for 40 minutes, three times a week, for five weeks.

Short Foot Exercise: Participants will sit with hips, knees, and ankles at 90 degrees, feet flat on the floor. They will pull their toes toward the heel to elevate the medial longitudinal arch, hold for 5 seconds, and relax. This will be repeated 15 times.

Towel Curl Exercise: Participants will sit with hips, knees, and ankles at 90 degrees, feet flat on the floor, with a towel placed under their feet. They will use their toes to gather the towel and then flatten it. This will be repeated 15 times.

Big Toe Press Exercise: Participants will press the big toe to the ground while lifting the other four toes, hold for 5 seconds, and repeat 15 times.

Toe Splay Exercise: Participants will sit with hips, knees, and ankles at 90 degrees, feet flat on the floor. They will spread the big toe and other toes apart, hold for 5 seconds, and repeat 15 times.

Calf Raise to Big Toe Press Exercise: Participants will stand barefoot on the edge of a step, lower their heels below the step level, rise onto their toes, and press onto the big toe, holding for 5 seconds. This will be repeated 15 times.

Leg Swings Exercise: Participants will stand barefoot on the affected foot, pulling the toes toward the heel to create an arch. The other leg will swing forward, backward, and side-to-side in small ranges of motion 15 times each.

Backward Tandem Walk Exercise: Participants will walk backward in a straight line, placing the heel of one foot directly in front of the toes of the other foot without deviating from the line.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25 to 60 years who have been diagnosed with plantar fasciitis by a physician specializing in physical medicine and rehabilitation or an orthopedic specialist.
* Heel pain localized to the medial calcaneal tubercle, persisting for three months or longer.
* Pain that worsens with the first steps taken in the morning or after periods of rest.

Exclusion Criteria:

* Individuals who have undergone foot or ankle surgery.
* Individuals with a history of chronic or active infection in the treatment area.
* Individuals with Type 1 or Type 2 Diabetes Mellitus, systemic inflammatory arthritis, cancer, active tuberculosis, or a history of neurological or vascular diseases.
* Individuals who have undergone conservative treatment including nonsteroidal anti-inflammatory drugs for 6 months with no significant improvement.
* Patients with numbness or tingling in the lower extremity, with or without provocation, or those with undiagnosed pain.
* Pregnancy.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only individuals who self-identify as female/male are eligible to participate.
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain | through study completion, an average of 6 months.
  The digital algometer is a pressure sensor used to measure pain thresholds by applying pressure to a specific point. In plantar fasciitis, it will assess foot sensitivity by measuring the pain threshold at the most painful area, especially the heel. Pressure is applied until pain is felt, and the recorded value indicates the threshold.
  The Visual Analog Scale (VAS) will evaluate heel pain by asking participants to mark their pain level on a 10 cm scale, where 0 means no pain and 10 signifies severe pain, based on their experience over the past week.
Medial longitudinal arc level | through study completion, an average of 6 months.
  The Navicular Drop Test will be used to assess participants' MLA height. Before measurements, the navicular tubercle will be marked while the individual stands barefoot. First, the distance between the navicular tubercle and the ground will be measured in millimeters while seated with the foot unloaded. Then, the individual will stand and bear full weight, and the new distance will be recorded. The difference between these two measurements will be calculated. Results will be classified as increased supination (<5mm), neutral foot (5-9mm), and increased pronation (>9mm).
Muscle strength | through study completion, an average of 6 months.
  The Kinvent K-Force digital device will be used for muscle strength measurement. Individuals with PF will lie in a supine position. For dorsiflexor strength measurement, the dynamometer will be placed on the upper metatarsal region, and for plantar flexors, it will be placed on the plantar metatarsal region. Participants will be asked to push against the dynamometer with maximum force, and the results will be recorded.
Quadriceps angle | through study completion, an average of 6 months.
  Changes in foot structure increase the Q angle, leading to genu valgum in the knee and pronation in the foot. Due to the tibia-talus relationship, foot pronation causes tibial internal rotation.
  Q angle measurement will be done using a plastic goniometer. Individuals with PF will lie supine with extended knees. The pivot point will be placed at the patella center. The movable arm will point to the anterior superior iliac spine, while the fixed arm will align with the tibial tuberosity. The angle between them will represent the Q angle

SECONDARY OUTCOMES:
Foot posture index | through study completion, an average of 6 months.
  Foot posture will be assessed using the Foot Posture Index (FPI). Individuals with PF will stand in a relaxed position, looking forward, with arms at their sides, maintaining body alignment.
  FPI includes six clinical criteria:
  * Talar head palpation
  * Curvatures above and below the lateral malleolus
  * Calcaneal inversion/eversion
  * Bulging in the talonavicular joint
  * MLA structure
  * Forefoot abduction/adduction relative to the rearfoot
  Each criterion is scored from -2 to +2, and the total score is recorded. A score of 0 indicates a neutral foot, positive values indicate pronation, and negative values indicate supination.
Foot function index | through study completion, an average of 6 months.
  The Foot Function Index (FFI) assesses foot pain, disability, and activity limitation through 23 items in three subcategories.
  The pain subscale measures foot pain levels in various situations. The disability subscale determines the difficulty of performing functional activities due to foot problems. The activity limitation subscale evaluates restrictions caused by foot issues.
  Patients will score all items based on their foot condition over the past week.

CONTACTS AND LOCATIONS:
Locations (1):
- Mudanya University, Bursa, Bursa, Turkey (Türkiye)